CLINICAL TRIAL: NCT03658681
Title: Fat Quality and Blood Glucose
Brief Title: Effect of Fat Quality on Glycemic Regulation and Gut Microbiota After a Short-time Intervention in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Mills DA (Industry); Nofima (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200642
Record Dates: First submitted 2018-06-06; First posted 2018-09-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2019-12

CONDITIONS: Postprandial Blood Glucose; Gut Microbiota; Satiety
Keywords: Fat quality; Blood glucose; Gut microbiota; Satiety; Dietary intervention

STUDY DESIGN:
Intervention Model Description: Intervention with cross-over design. Two test meals will be tested.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test meal 1: Saturated fat 14.9 E% (Experimental): Test meal with saturated fat 14.9 E%
  Interventions: Other: Saturated fat 14.9 E%
- Test meal 2: Polyunsaturated fat 13.6 E% (Experimental): Test meal with polyunsaturated fat 13,6 E%
  Interventions: Other: Polyunsaturated fat 13.6 E%

INTERVENTIONS:
Other: Saturated fat 14.9 E% — Dietary cross-over study with saturated fat
  Arms: Test meal 1: Saturated fat 14.9 E%
Other: Polyunsaturated fat 13.6 E% — Dietary cross-over study with polyunsaturated fat
  Arms: Test meal 2: Polyunsaturated fat 13.6 E%

SUMMARY:
The overall aim is to investigate effects of saturated versus polyunsaturated fat on glycemic regulation and satiety in a postprandial study with healthy individuals. The potential effects will be related to changes in gut microbiota, the circulating levels of short chain fatty acids, inflammation and gene expression in peripheral mononuclear blood cells.

DETAILED DESCRIPTION:
The intervention study will have a randomized, double blinded, cross-over design with different test meals consisting of saturated or polyunsaturated fat. The amount of fat will be identical in the test meals, but the fat quality will vary. The test meals are in the form of muffin and spread.

All participants will consume two muffins and minimum 20 g of spread a day for three consecutive days, consisting of either a high proportion of saturated fat or a high proportion of polyunsaturated fat. At day one (visit 1 and 3) and day four (visit 2 and 4) of the intervention week, the participants will perform a postprandial glucose test (OGTT, 75 g glucose in 100 ml water) at Oslo Metropolitan University. Blood samples will be taken before and at different time points after the glucose test. One week prior to the intervention week and during "wash-out" (11 days), the participants will consume the control products which are high in saturated fat.

At the screening visit (visit 0) the participants will be asked to limit the intake of dietary fat and fiber from oat and barley one week prior to visit 1 and during the study. Otherwise, participants will be asked not to change their diet and exercise habits during the study period. Individuals fulfilling the inclusion criteria will also be invited to participate in a cross-sectional study for investigating the gut microbiota in a healthy population.

An OGTT will be performed at visit 1, 2, 3 and 4.

The participants will receive test meals after screening and before visit 1, 2, and 3.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18,5 and 27 kg/m2
* Fasting plasma glucose ≤ 6.1 mmol/l

Exclusion Criteria:

* Chronic metabolic diseases such as diabetes type 1 and 2, coronary heart disease and cancer the last 6 months.
* Intestinal diseases such as chron's disease, ulcerative colitis and irritable bowel syndrome.
* Food allergy and intolerances towards grain and dairy products.
* Pregnant and lactating
* Smokers
* Fasting blood glucose ≥ 6.1 mmol/L
* BMI <18,5 and >27 kg/m2
* Planned weight reduction and or ± 5% weight change over the past three months.
* Use of antibiotics last 3 months before study entry and during the study period
* Use of probiotics the last month before study entry and during the study period
* Blood donor last 2 months before study entry and or during the study period
* Not willing to end the use of dietary supplements, including probiotic products, fish oil etc. four weeks prior to study entry and throughout the study period
* Alcohol consumption > 40g / day
* Hormone treatments (except contraceptives)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose response measured in capillary blood | Change from baseline at day 4
  Blood glucose response after oral glucose tolerance test (OGTT) measured in Finger-prick capillary blood samples
Serum Insulin response measured in venous blood samples | Change from baseline at day 4
  Serum Insulin response after OGTT measured in venous blood samples

SECONDARY OUTCOMES:
Hydrogen breath response measured in expired air | Change from baseline at day 4
  Hydrogen breath response after OGTT measured in expired air by Gastroanalyzer
Free fatty acids | Change from baseline at day 4
  Plasma free fatty acids are measured after intake of test meals
Microbiota analyses in feces | Change from baseline at day 4
  Microbiota analyses in feces are measured before and after intake of test meals. Change in microbiota will be analysed
Serum triglyceride response | Change from baseline at day 4
  Triglyceride response are measured are measured after OGTT
Serum cholesterol | Change from baseline at day 4
  Serum cholesterol are measured fasting after intake of test meals
Hunger and satiety hormones (e.g. GLP2, PYY) | Change from baseline at day 4
  The response in hunger and satiety hormones after OGTT
Inflammatory markers (e.g. CRP) | Change from baseline at day 4
  Response in Inflammatory markers are measured after OGTT
mRNA analyses in PBMC | Change from baseline at day 4
  PBMC are collected before and after OGTT. The change in mRNA level will be analyzed
Quantitative assessment of metabolites in urine | Change from baseline at day 4
  Morning urine are collected before and after intake of test meals. Metabolites in urine will be quantified using UHPLC-qTOF-MS. Change in metabolites before and after test meals will be analyzed
Quantitative assessment of metabolites in plasma | Change from baseline at day 4
  Plasma for metabolome analyses are collected after intake of test meals. Metabolites in plasma will be quantified using UHPLC-qTOF-MS
Visual analogue scale (VAS) | Change from baseline at day 4
  Subjective hunger and satiety after OGTT and will be measured on a 100 mm horizontal line. Marks towards right end on line indicates strong sensation for hunger and satiety, whereas marks towards left end indicates opposite sensation. The distance from left border of line to the mark indicates subjective sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Telle-Hansen, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Telle-Hansen VH, Gaundal L, Bastani N, Rud I, Byfuglien MG, Gjovaag T, Retterstol K, Holven KB, Ulven SM, Myhrstad MCW. Replacing saturated fatty acids with polyunsaturated fatty acids increases the abundance of Lachnospiraceae and is associated with reduced total cholesterol levels-a randomized controlled trial in healthy individuals. Lipids Health Dis. 2022 Sep 26;21(1):92. doi: 10.1186/s12944-022-01702-1. PMID 36163070